CLINICAL TRIAL: NCT01605994
Title: Placebo-Controlled, Multiple Ascending-Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BMS-933043
Brief Title: Multiple Ascending-Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BMS-933043 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CN171-002
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Adult Normals
MeSH Terms: interventions — BMS-933043

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- Panel 1:BMS-933043(2mg)/Placebo+Antacid Buffer Solution (Experimental): BMS-933043 2 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- Panel 2:BMS-933043(5mg)/Placebo+Antacid Buffer Solution (Experimental): BMS-933043 5 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- Panel 3:BMS-933043(10mg)/Placebo+Antacid Buffer Solution (Experimental): BMS-933043 10 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- Panel 4:BMS-933043(25mg)/Placebo+Antacid Buffer Solution (Experimental): BMS-933043 25 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- Panel 5:BMS-933043(50mg)/Placebo+Antacid Buffer Solution (Experimental): BMS-933043 50 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  CSF sampling required
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- Panel 6:BMS-933043(100mg)/Placebo+Antacid Buffer Solution (Experimental): BMS-933043 100 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- Panel 7:BMS-933043(200mg)/Placebo+Antacid Buffer Solution (Experimental): BMS-933043 200 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- Panel 8:BMS-933043(25mg)/Placebo+Antacid Buffer Predose (Experimental): MAD Phase: Japanese Subjects. Cerebrospinal fluid (CSF) sampling not required
  BMS-933043 25 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- Panel 9:BMS-933043(200mg)/Placebo+Antacid Buffer Predose (Experimental): Japanese Subjects. CSF sampling not required.
  BMS-933043 200 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- Panel 10:BMS-933043(350mg)/Placebo+Antacid Buffer Predose (Experimental): BMS-933043 350 mg solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution
- CSF Panel:BMS-933043(MTD)/Placebo+Antacid Buffer Predose (Experimental): If Panel 5 does not run. CSF Sampling at steady state
  BMS-933043 maximum tolerated dose (MTD), solution by mouth twice daily for 10 days
  OR
  Placebo matching with BMS-933043 0 mg solution by mouth twice daily for 10 days
  Antacid Buffer Predose 150 mL solution by mouth twice daily for 10 days
  Interventions: Drug: BMS-933043; Drug: Placebo matching with BMS-933043; Drug: Antacid Buffer Predose Solution

INTERVENTIONS:
Drug: BMS-933043
Drug: Placebo matching with BMS-933043
Drug: Antacid Buffer Predose Solution

SUMMARY:
Includes a placebo-controlled sequential, ascending multiple-dose panels (10 panels, 8 ascending doses, and 2 fixed Japanese Panels exploring safety, tolerability, and Pharmacokinetic (PK) measures

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal medical history, physical examination, ECGs and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 30 kg/m2, inclusive. BMI = weight (kg)/ [height (m)]2
* Normal Neurological Exam (LP subjects only: to rule out focal CNS lesions that would render LP unsafe)
* Men and women, ages 18 to 55 years, inclusive.
* Women who are not of childbearing potential (WOCBP) [ie, who are postmenopausal or surgically sterile] and men
* Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
* Women must not be breastfeeding
* Sexually active fertile men must use effective birth control if their partners are WOCBP throughout the study and for 90 days after last dose

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study drug administration) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery that could impact upon the absorption of study drug
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks of study drug administration
* Blood transfusion within 4 weeks of study drug administration
* Inability to tolerate oral medication
* Inability to be venipunctured and/or tolerate venous access
* Smoking more than 1 cigarette/cigar per week, within 3 months prior to screening
* Regular daily use of nicotine products or Varenicline (Chantix® or Champix®) within 3 months prior to screening
* Recent (within 6 months of study drug administration) drug or alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders (4th Edition) [DSM IV], Diagnostic Criteria for Drug and Alcohol Abuse
* History of cardiac arrhythmias, or palpitations associated with presyncope or syncope or history of unexplained syncope

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple oral doses of BMS-933043 in healthy subjects measured by AEs, Vital signs, clinical laboratory test results, physical examination findings, neurological examination findings and electrocardiogram (ECG) parameters | Up to Day 26 of Follow-up
  AEs = Adverse Events

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12
  PK of BMS-933043, BMS-941651, BMS-972869 and BMS-610999 will be derived from plasma concentration versus time and urinary excretion data
Time of maximum observed plasma concentration (Tmax) | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12
  PK of BMS-933043, BMS-941651, BMS-972869 and BMS-610999 will be derived from plasma concentration versus time and urinary excretion data
Area under the concentration-time curve in one dosing interval [AUC(TAU)] | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12
  PK of BMS-933043, BMS-941651, BMS-972869 and BMS-610999 will be derived from plasma concentration versus time and urinary excretion data
Plasma half-life (T-HALF) | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12
  PK of BMS-933043, BMS-941651, BMS-972869 and BMS-610999 will be derived from plasma concentration versus time and urinary excretion data
Trough observed plasma concentration (Cmin) between dose interval | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12
  PK of BMS-933043, BMS-941651, BMS-972869 and BMS-610999 will be derived from plasma concentration versus time and urinary excretion data
Volume of distribution at steady-state (VSS/F) of BMS-933043 | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12
  PK of BMS-933043 will be derived from plasma concentration versus time and urinary excretion data
Accumulation index (AI): ratio of AUC(TAU) at steady-state to AUC(TAU) after the first dose | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12
  PK of BMS-933043, BMS-941651, BMS-972869 and BMS-610999 will be derived from plasma concentration versus time and urinary excretion data
Ratio of metabolite AUC(TAU) to parent AUC(TAU), corrected for molecular weight [MR AUC(tau)] | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12
  PK of BMS-933043, BMS-941651, BMS-972869 and BMS-610999 will be derived from plasma concentration versus time and urinary excretion data
Ratio of metabolite Cmax to parent Cmax, corrected for molecular weight [MR Cmax] | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12
  PK of BMS-933043, BMS-941651, BMS-972869 and BMS-610999 will be derived from plasma concentration versus time and urinary excretion data
CSF penetration of BMS-933043 | Day 8
  Cerebral Spinal Fluid (CSF) will be analyzed for drug levels to confirm adequate central nervous system (CNS) penetration (>2 nM is required) and to estimate the brain/plasma ratio in humans
Effect of BMS-933043 on ECG intervals and to explore the relationship between plasma exposure and ECG intervals | Baseline (Day -2), Day 1, Day 6 and Day 10
  The effects of BMS-933043 on ECG parameters (heart rate, QTcF, PR, and QRS) will be explored graphically and by summary statistics. Absolute levels, as well as changes from baseline, will be summarized and plotted versus time by treatment and day for each ECG parameter. Frequency distributions for subjects' maximum values will be provided by treatment. The relationships between ECG parameters and BMS-933043 concentrations may be explored using scatter plots and the relationship between the change from baseline in QTcF and the BMS-933043 concentration may be estimated
Safety and tolerability of multiple oral doses of BMS-9333043 in Japanese healthy subjects is measured by AEs, Vital signs, clinical laboratory test results, physical examination findings, neurological examination findings and ECG parameters | Up to 6 months
Effect of ethnicity (Japanese versus non-Japanese) on PK of BMS-933043 will be assessed graphically and by point estimates and 90% confidence intervals for geometric mean ratio for Cmax using data from subjects receiving the same dose of BMS-933043 | Day 1, Day 3, Day 6, Day 9, Day 10, Day 11 and Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Clinilabs, Inc., New York, New York, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx